CLINICAL TRIAL: NCT01294826
Title: Phase IB With Expansion of Patients at the MTD Study of AUY922 and Cetuximab in Patients With KRAS Wild-Type Metastatic Colorectal Cancer
Brief Title: Study of AUY922 and Cetuximab in Patients With KRAS Wild-Type Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922AUS06T
Record Dates: First submitted 2011-02-08; First posted 2011-02-14 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
Keywords: Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Cetuximab; HSP90 Heat-Shock Proteins; EGFR protein, human
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AUY922 plus Cetuximab (Experimental)
  Interventions: Drug: AUY922; Drug: Cetuximab

INTERVENTIONS:
Drug: AUY922 — Weekly intravenous infusion on Day 1, 8, 15 and 22 of each 28 day cycle until unacceptable toxicity develops or disease progression. A minimum of 3 patients will be enrolled into each cohort. The anticipated dose escalation sequence of AUY922 is 40, 55, and 70 mg/m2 will be used.
Drug: Cetuximab — Cetuximab will be administered after each AUY922 infusion, intravenously on Day 1, 8, 15 and 22 of each 28 day cycle until unacceptable toxicity develops or disease progression.

SUMMARY:
The study will determine the maximum tolerated dose (MTD) of AUY922 given in combination with cetuximab in previously treated patients with KRAS wild-type metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal cancer
* KRAS wild type metastatic colorectal cancer
* Progression of disease on at least 2 prior therapy to have included 5FU, or oxaliplatin or bevacizumab or irinotecan
* Prior treatment with cetuximab is allowed (full dose tolerated), provided that the patient never required a dose reduction due to toxicities
* Must have at least one measurable lesion
* Must be 18 years of age or older
* ECOG performance status 0-1
* Life expectancy must be greater than 12 weeks
* For women of childbearing potential, a negative pregnancy blood test must be obtained less than 3 days prior to the first AUY922 infusion

Exclusion Criteria:

* Colorectal cancer with a KRAS mutation or in which the KRAS genotype status is unknown
* Metastasis to the CNS
* Prior treatment with any Hsp90 inhibitor compounds
* Patients who received systemic anti-cancer treatment prior to the first dose of AUY922 within the following time frames:

  * Radiotherapy, conventional chemotherapy: within 2 weeks
  * Palliative radiotherapy: within 2 weeks
  * Nitrosoureas, monoclonal antibodies, such as trastuzumab and mitomycin: within 6 weeks
  * Any continuous-dosing (i.e. daily dosing, every-other-day dosing, Monday-Wednesday-Friday dosing, weekly etc.) of systemic anti-cancer treatment for which the recover period is not known, or investigational drugs (i.e. targeted agents) within a duration of ≤ 5 half lives of the agent and their active metabolites (if any)
* Treatment of therapeutic doses of coumadin-type anticoagulants. [Maximum daily dose of 2mg, for line patency permitted]
* Known sensitivity to cetuximab
* Unresolved ≥ grade 1 diarrhea
* Malignant ascites that require invasive treatment
* Concurrent medications that are substrates, inhibitors or inducers of CYP3A4, CYP2C8, CYP2C9 and CYP2C19 and cannot be switched or discontinued or switched to an alternative drug prior to commencing AUY922 dosing need special consideration on a case by case basis
* Major surgery ≤ 2 weeks prior to randomization or who have not recovered from such therapy
* Impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | 1 cycle (1 cycle = 28 days)

SECONDARY OUTCOMES:
Patient response rate to the AUY922. | After 2 years
Time to tumor progression following treatment with AUY922. | After 2 years
Overall survival of patients treated with AUY922. | After 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gold, MD, Principal Investigator — Swedish Medical Center Cancer Institute
Locations (1):
- Swedish Medical Center Cancer Institute, Seattle, Washington, United States